CLINICAL TRIAL: NCT05557136
Title: The Effectiveness of Polyether-Ether-Ketone (PEEK) as a Fixed Retainer Compared to Multistranded Stainless Steel Wires: A Randomized Clinical Trial
Brief Title: Effectiveness of PEEK Fixed Retainer
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Esraa Salman Jasim (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Sponsor-Investigator, Esraa Salman Jasim, Assist.Prof., University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 621422
Record Dates: First submitted 2022-09-02; First posted 2022-09-27 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Retention
Keywords: Retention; Stability; Periodontal indices; Fixed retainer; PEEK
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multistranded stainless steel fixed retainer (Experimental): Multistranded stainless steel fixed retainer is used for lower anterior teeth (canine to canine) to maintain the stability of teeth after completion of orthodontic treatment
  Interventions: Device: Multistranded stainless steel fixed retainer
- Polyether-Ether-Ketone (PEEK) fixed retainer (Experimental): Polyether-Ether-Ketone (PEEK) fixed retainer is used for lower anterior teeth (canine to canine) to maintain the stability of teeth after completion of orthodontic treatment
  Interventions: Device: Polyether-Ether-Ketone (PEEK) fixed retainer

INTERVENTIONS:
Device: Multistranded stainless steel fixed retainer — Multistranded stainless steel fixed retainer is used for orthodontic patient after completion of orthodontic treatment to achieve stability of alignment.
  Arms: Multistranded stainless steel fixed retainer
Device: Polyether-Ether-Ketone (PEEK) fixed retainer — Polyether-Ether-Ketone (PEEK) fixed retainer is used for orthodontic patient after completion of orthodontic treatment to achieve stability of alignment.
  Arms: Polyether-Ether-Ketone (PEEK) fixed retainer

SUMMARY:
A randomized clinical trial is set out to compare the effectiveness of two types of fixed retainer (multistranded stainless steel and PEEK types) in maintaining the stability of lower anterior teeth with less failure rate.

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two arms parallel group. The patients will be randomly divided into two groups, group one: multistranded stainless steel fixed retainer will be used while, and group two PEEK fixed retainer will be used. An intra-oral scan, intra-oral swap and periodontal indices will be taken before starting the treatment (T0), after one month (T1), after 3 months (T2), and after 6 months (T3). Patient perception concerning the fixed retainer will be taken for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 17-32 years.
* Patients with a score of 0-0.5 on Little's irregularity index in the lower arch.
* Patients treated with the pre-adjusted orthodontic appliance (both Extraction and non-extraction cases).
* Patients who have healthy periodontal condition

Exclusion Criteria:

* Patients treated with rapid maxillary expansion or surgically assisted rapid maxillary expansion.
* Patients with a cleft lip / and or palate.
* Patients with a deep overbite and traumatic parafunctional habits such as bruxism and clenching.
* Patients with carious, restored, fractured, or missing lower anterior teeth.
* Patients with medical health problems that may influence gingival health like uncontrolled type II diabetic patient, patients with hormonal disturbances or systemic drug administration that effect on oral health.
* Smokers

Ages: 12 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Stability of lower anterior teeth | T0 is the stating of retention, T1 after one month, T2 after 3 months and T3 after 6 month
  The effectiveness of PEEK retainers as compared to a dead-soft multi-stranded stainless-steel wire in maintaining alignment of the lower anterior teeth in terms of Little's irregularity index.

SECONDARY OUTCOMES:
Failure rate | T0 is the stating of retention, T1 after one month, T2 after 3 months and T3 after 6 month
  how many times the retainer needed to be replaced or repaired
Periodontal health status | T0 is the stating of retention, T1 after one month, T2 after 3 months and T3 after 6 month
  The effect of fixed retainer on the periodontal health is measured by oral hygiene indices
Patient satisfaction | At T1 after one month and T3 after 6 month
  Patient satisfaction concerning esthetics, speech and comfort is obtain by questionnaire.
Biohostability | T0 is the stating of retention, T1 after one month, T2 after 3 months and T3 after 6 month
  studying the microbial colonization on the retainer wire by using oral swap of fixed retainer and measure total bacterial count (Aerobic and Facultative Anaerobic) on Blood agar, Total streptococcus count and total lactobacillus count on selective media

CONTACTS AND LOCATIONS:
Overall Officials: Ammar S Kadhum, Study Director — University of Baghdad
Locations (1):
- Esraa S Jasim, Baghdad, Baghdad, Bab Al-Moadham, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jasim ES, Kadhum AS. Poly-Ether-Ether-Ketone versus dead-soft coaxial bonded retainers: a randomized clinical trial. Part 2: periodontal health and microbial biofilm assessment. Eur J Orthod. 2024 Oct 1;46(5):cjae048. doi: 10.1093/ejo/cjae048. PMID 39312715
- [Derived] Jasim ES, Kadhum AS. Poly-ether-ether-ketone (PEEK) versus dead-soft coaxial bonded retainers: a randomized clinical trial. Part 1. Stability, retainer failure, and participant satisfaction. Eur J Orthod. 2024 Oct 1;46(5):cjae044. doi: 10.1093/ejo/cjae044. PMID 39206494